CLINICAL TRIAL: NCT02895555
Title: RCT Comparing i-FACTOR and Allograft in Spinal Fusion Surgery
Brief Title: The Clinical Effect of i-FACTOR® Versus Allograft in Non-instrumented Posterolateral Fusion The IVANOS-study
Acronym: IVANOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spine Centre of Southern Denmark (Other)
Collaborators: Ortotech (Unknown); CeraPedics, Inc (Industry)
Responsible Party: Principal Investigator, Karen Højmark Hansen, Research coordinator, Spine Centre of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20120012; 20180146 (Other: Ethics comitee)
Record Dates: First submitted 2013-06-24; First posted 2016-09-09 (Estimated); Last update posted 2024-04-19 (Actual); Status verified 2018-11

CONDITIONS: Spinal Stenosis; Low Back Pain
Keywords: Oswestry disability index (ODI)
MeSH Terms: conditions — Spinal Stenosis; Low Back Pain | interventions — Fibrinogen; Cyclin-Dependent Kinase Inhibitor p15; Transplantation, Homologous

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Allograft group, standard treatment (Active Comparator): Control group, standard treatment. Approx 50 g pr level fused.
  Interventions: Procedure: Allograft
- i-FACTOR (Experimental): i-FACTOR putty in the operation site. Fda approved. Approx 5 ml pr level fused.
  Interventions: Procedure: i-FACTOR

INTERVENTIONS:
Procedure: i-FACTOR — Between 5-10 CC i-FACTOR putty mixed with local harvested autograft pr level spondylodesis compared to 30 grams of allograft pr level mixed with local harvested allograft.
  Other Names: P15
  Arms: i-FACTOR
Procedure: Allograft — Approx 50 g of allograft bone in the fused site
  Arms: Allograft group, standard treatment

SUMMARY:
The average life expectancy in Denmark is increasing resulting in an increasing part of the population having age-related disease, ex lumbar spinal stenosis (LSS). LSS causes constriction of the nerves in the lumbar spine resulting in pain in the legs and lower back, especially when standing and walking, known as neurogenic claudicatio(Goh KJ FAU - Khalifa et al.). LSS occurs in a combination of degenerative changes in the lower back, including hypertrophy of the ligamentum flavum, arthrosis of the facet joints and bulging of the disc.

Current treatment of LSS is varied ranging from non-operative conservative treatment to operation.

Operative intervention shows very good results according to physical ability and pain(Christensen FB et al.;Hee HT and Wong;McGregor AH FAU - Hughes and Hughes;Xu et al.), but the most optimal treatment is still debated. Nevertheless, a decompression and, if needed, a spinal fusion is recommended.

The investigators want to se whether i-FACTOR improves clinical outcomes compared to using allograft in spinal fusion in the elderly, and thereby find an improved methods operating this difficult patient population.

The hypothesis is, that there is no difference in clinical outcomes whether you use i-FACTOR or allograft i non-instrumented spinal fusion surgery in patients with spinal stenosis due to degenerative listhesis.

DETAILED DESCRIPTION:
Se above

ELIGIBILITY:
Inclusion Criteria:

1. Spinal stenosis, listhesis grade 1-2 (>3 mm), facet joint arthrosis and flavum hypertrophia verified by a mr-scan and x-ray including maximally 2 levels ranging from L1-S1.
2. A score of 6 and more on Konno´s "History of Examination Characteristic".
3. Signed informed content.

Exclusion Criteria:

1. Any disease demanding obligate thromboprophylaxis treatment, including mechanical valve, (DVT with cancer/thrombophilia, AMI, apoplexia cerebri, TCI, valve-operation)< 3 months, coronar metal stent < 6 weeks and coronar drug eluted/coated stent < 12 months.
2. Atrial fibrillation and one of the following: Mitral stenosis, valve prothesis and apoplexia cerebri/TCI.
3. Atrial fibrillation and two of the following: Heart insufficient, HT, DM, age > 75 years, EF < 35 %.
4. Known cancer in the axial skeleton.
5. Ongoing chemotherapy.
6. Fracture i the lower back within a year prior to inclusion.
7. Reduced distance of walking due to non-spinal related causes.
8. Candidate for more than two-level intervention.
9. Dementia assessed by the MMSE
10. ASA 3+4
11. Age below 60 years.
12. Missed 3 months of conservative treatment without success
13. The use of steroids and bisphosphonates.
14. Prior radiotherapy to the lower back.
15. Haematologic disease. -

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Oswestry disability index | At 60 months
  questionnaire

SECONDARY OUTCOMES:
Dallas pain questionnaire | At 24 months
  questionnaire
Walking distance | At 24 months
  measuring distance
EQ5D | At 60 months
  questionnaire
SF-36 | At 60 months
  questionnaire
Fusion status yes/no | At 60 months
  Obtained by CT-scan

CONTACTS AND LOCATIONS:
Overall Officials: Mikkel Andersen, MD, Principal Investigator — Department of spine surgery of Southern Denmark
Locations (1):
- Middelfart spine surgery research department, Middelfart, Denmark

IPD SHARING:
Plan to Share IPD: Undecided